CLINICAL TRIAL: NCT00078585
Title: A Phase II Randomized, Double Blind, Controlled Study to Evaluate the Safety and Efficacy of PROSTVAC®-VF/TRICOM™ in Combination With GM-CSF in Patients With Androgen-Independent Adenocarcinoma of the Prostate
Brief Title: PROSTVAC®-VF/TRICOM™ Vaccine for the Treatment of Metastatic Prostate Cancer After Failing Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: Therion Biologics Corporation (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: TBC-PRO-002; NCT00081120 (obsolete NCT alias)
Record Dates: First submitted 2004-03-01; First posted 2004-03-03 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Biological: PROSTVAC®-VF/TRICOM™

SUMMARY:
PROSTVAC-VF is an investigational cancer vaccine. The vaccine is based on the theory that the immune system can be taught to fight cancer by directing the immune system to attack specific targets found on cancer cells. These targets are called Tumor Associated Antigens, or TAA's. This trial will help determine if this vaccine can help fight cancer.

This multi-center, double-blind, randomized, empty vector-controlled trial is designed to evaluate the safety and efficacy of PROSTVAC-VF/TRICOM co-administered with GM-CSF versus the empty viral vector co-administered with placebo in the treatment of patients with androgen-independent prostate cancer (AIPC).

All patients will be required to sign an informed consent prior to the performance of any on-study procedures. Patients will be screened for eligibility within 14 days prior to vaccine administration. Patients who meet all inclusion and exclusion criteria will be centrally randomized into the study and will receive a unique patient identification number and a blinded treatment assignment. The ratio of active treatment to empty vector control (placebo) is 2:1.

ELIGIBILITY:
* Male patients > 18 years of age who have been vaccinated against smallpox;
* Histological confirmation of adenocarcinoma of the prostate with evidence of metastatic disease including either of the following: Lymph node metastasis measurable by CT and/or Bone metastasis evaluable by bone scan;
* Despite hormone therapy, there is evidence of two consecutive increases in PSA (Prostate Specific Antigen);
* Gleason Score of 7 or lower at initial diagnosis.

Please note that there are additional eligibility criteria that you must meet to qualify.

If you do qualify to participate, study personnel will explain the trial in detail and answer any questions you may have. You can then decide whether or not you wish to participate. If you do not qualify for the trial, study personnel will explain the reasons.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2003-11; Primary Completion 2006-01-04 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Schuetz, MD, Study Director — Therion Biologics Corporation; Philip W Kanthoff, MD, Principal Investigator — Dana-Faber Cancer Institut
Locations (47):
- United States (47):
  - Urology Centers of Alabama, Homewood, Alabama
  - Alaska Clinical Research Center, Anchorage, Alaska
  - Urology Associates of Central California, Fresno, California
  - San Diego Urology Center, La Mesa, California
  - Loma Linda University, Loma Linda, California
  - Atlantic Urology Medical Group, Long Beach, California
  - Pacific Clinical Research, Santa Monica, California
  - Western Clinical Research, Inc., Torrance, California
  - UCHSC Anschutz Cancer Pavilion, Aurora, Colorado
  - Connecticut Clinical Research Center, Waterbury, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia
  - South Florida Medical Research, Aventura, Florida
  - Advanced Research Institute, New Port Richey, Florida
  - Midtown Urology, Atlanta, Georgia
  - North Idaho Urology, Coeur d'Alene, Idaho
  - Prairie Medical Associates, Ltd., Chicago, Illinois
  - Medical and Surgical Specialists, Galesburg, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Carle Clinic Cancer Center, Urbana, Illinois
  - Metropolitan Urology, Jeffersonville, Indiana
  - Urologic Associates, PC, Davenport, Iowa
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Lawrenceville Urology, Lawrenceville, New Jersey
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Urology Group of New Mexico, Albuquerque, New Mexico
  - The Urological Institute of Northeastern New York, Albany, New York
  - AccuMed Research Associates, Garden City, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - Nyack Hospital, Nyack, New York
  - The Urology Center, Greensboro, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Charleston Cancer Center, Charleston, South Carolina
  - Urology Associates Clinical Research, Nashville, Tennessee
  - Arlington Cancer Center, Arlington, Texas
  - Urology Clinic of North Texas, PA, Dallas, Texas
  - Texas Cancer Center, Fort Worth, Texas
  - Texas Cancer Care, Weatherford, Texas
  - Salt Lake Research, Salt Lake City, Utah
  - University of Vermont, South Burlington, Vermont
  - Virginia Urology Center, Richmond, Virginia
  - McGuire Research Institute, Richmond, Virginia
  - Midwest Research Specialists, LLC, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Wyoming Research Foundation, Inc., Cheyenne, Wyoming

REFERENCES:
- [Result] Kantoff PW, Schuetz TJ, Blumenstein BA, Glode LM, Bilhartz DL, Wyand M, Manson K, Panicali DL, Laus R, Schlom J, Dahut WL, Arlen PM, Gulley JL, Godfrey WR. Overall survival analysis of a phase II randomized controlled trial of a Poxviral-based PSA-targeted immunotherapy in metastatic castration-resistant prostate cancer. J Clin Oncol. 2010 Mar 1;28(7):1099-105. doi: 10.1200/JCO.2009.25.0597. Epub 2010 Jan 25. PMID 20100959
- [Result] Kantoff PW, Gulley JL, Pico-Navarro C. Revised Overall Survival Analysis of a Phase II, Randomized, Double-Blind, Controlled Study of PROSTVAC in Men With Metastatic Castration-Resistant Prostate Cancer. J Clin Oncol. 2017 Jan;35(1):124-125. doi: 10.1200/JCO.2016.69.7748. Epub 2016 Sep 30. No abstract available. PMID 27646950